CLINICAL TRIAL: NCT05266144
Title: A Prospective Cohort Study of Atrial Fibrillation Patients Treated With Catheter Ablation
Brief Title: Atrial Fibrillation Patients Treated With Catheter Ablation
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-AF
Record Dates: First submitted 2022-02-13; First posted 2022-03-04 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation Recurrent
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will be used for biochemical parameter analysis, and atrial fibrillation patients with ventricular fibrosis will be selected for gene sequencing to explore the existence of underlying cardiomyopathy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- atrial fibrillation: Atrial fibrillation patients who underwent radiofrequency ablation in Peking Union Medical College Hospital.
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: radiofrequency ablation — Bilateral pulmonary vein isolation, a kind of radiofrequency ablation, is performed in atrial fibrillation patients for atrial arrhythmia therapy.

SUMMARY:
This is a single-center prospective observational cohort study of atrial fibrillation patients treated with radiofrequency ablation.

DETAILED DESCRIPTION:
The effect of radiofrequency therapy on the life quality and atrial function of atrial fibrillation patients will be assessed, through the multidimensional analysis of baseline clinical data, serological indicators of atrial fibrosis, echocardiography, cardiac magnetic resonance imaging, atrial potential mapping, life quality, and long-term ECG monitoring within 1 week after radiofrequency ablation. A predictive model for atrial fibrillation recurrence after ablation will be established. Based on the cross-sectional analysis of baseline data, the relationship between non-invasive assessment of atrial fibrosis (imaging and serology), atrial electrical activity, and atrial function will be analyzed as well, and atrial fibrillation patients with ventricular fibrosis will be selected for gene sequencing to explore the existence of underlying cardiomyopathy and provide data for further research.

ELIGIBILITY:
Inclusion Criteria:

* Non-valvular atrial fibrillation, including paroxysmal atrial fibrillation and persistent atrial fibrillation
* 18-80 years old
* The anteroposterior diameter of the left atrium is less than 50mm via TTE
* Patient meets the intervention criteria for bilateral pulmonary vein isolation after evaluation by electrophysiological specialists
* Patient consents to ablation treatment

Exclusion Criteria:

* Intra-atrial thrombus detected by TEE
* Hyperthyroidism
* Previous radiofrequency ablation for atrial fibrillation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive atrial fibrillation patients, who underwent catheter ablation in Peking Union Medical College Hospital, were enrolled. All patients went through bilateral pulmonary vein isolation under general or local anesthesia, and were regularly followed up at 3-month and 1-year after ablation.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence assessed by ECG, Holter reports and outpatient physicians | at 1-year follow-up after ablation
  Recurrence includes atrial fibrillation and atrial flutter. Recurrence features including pattern, duration, burden, etc. will be recorded.
All-cause mortality assessed by telephone follow-up or medical records | at 1-year follow-up after ablation
  Time and cause of death will be recorded.

SECONDARY OUTCOMES:
Improvement in life quality assessed by QOLSF36 Questionnaire | at 1-year follow-up after ablation
  Life quality will be assessed at baseline and 1-year FU. Improvement in life quality indicates that patients can benefit from the catheter ablation.
Improvement in left atrial function assessed by echocardiography | at 1-year follow-up after ablation
  Left atrial function will be assessed at baseline and 1-year FU. Improvement in atrial function indicates that ablation can restore atrial function.
Embolic events assessed by physicians and further examinations like ultrasound, MRI | at 1-year follow-up after ablation
  Embolism may be related to atrial fibrillation. Embolism will be assessed by physicians according to patients' symptoms and signs at clinic or by telephone. If a patient's clinical presentation indicates embolism, the patient will be further assessed by ultrasound, MRI, etc.
Hospitalization for heart failure, atrial fibrillation or atrial flutter | at 1-year follow-up after ablation
  Postoperative hospitalization indicate worse prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Quan Fang, M.D., Study Chair — Peking Union Medical College Hospital; Yongtai Liu, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Sun K, Qin X, Zhang D, Fang F, Wan R, Wang J, Yu J, Lai J, Yang D, Fan J, Cheng Z, Cheng K, Gao P, Zhang L, Deng H, Fang Q, Chen T, Liu Y. HFpEF correlated with better improvement of left atrial function in post-ablation patients with paroxysmal atrial fibrillation. Int J Cardiovasc Imaging. 2025 Apr;41(4):721-732. doi: 10.1007/s10554-025-03359-0. Epub 2025 Mar 1. PMID 40025277